CLINICAL TRIAL: NCT05587049
Title: Effectiveness and Safety of Venetoclax in Combination With Azacitidine in Patients With Acute Myeloid Leukemia in Real Life Clinical Practice
Brief Title: A Study to Assess Change in Disease State in Adult Participants With Acute Myeloid Leukemia (AML) Receiving Oral Venetoclax Tablets in Combination With Subcutaneously (SC) or Intravenously (IV) Injected Azacitidine in Colombia
Acronym: ESVECO
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-469
Record Dates: First submitted 2022-10-18; First posted 2022-10-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Venetoclax; Venclexta; Venclyxto; Azacitidine; ABT-199; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax + Azacitidine Participants: Participants treated with venetoclax in combination with azacitidine in accordance with approved local label.

SUMMARY:
Acute myeloid leukemia (AML) is a cancer of the blood and bone marrow and is the most common acute leukemia in adults. This study will evaluate how well venetoclax in combination with azacitidine works to treat AML in adult participants in Colombia.

Venetoclax in combination with azacytidine is approved to treat Acute myeloid leukemia (AML). All study participants will receive venetoclax in combination with azacitidine as prescribed by their study doctor in accordance with approved local label. Adult participants with a new diagnosis of AML will be enrolled. Around 70 participants will be enrolled in the study in Colombia.

Participants will receive venetoclax tablets to be taken by mouth in combination with azacitidine given by subcutaneous (SC) or intravenous (IV) injection according to the approved local label. The duration of the study is approximately 36 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute myeloid leukemia (AML) defined as participants that have histological confirmation of AML (de novo, secondary) by World Health Organization (WHO) criteria, and have not received any prior treatment for AML.
* Ineligible to intensive chemotherapy due to >=75 years of age; or >=18 to 74 years who have comorbidities that preclude use of intensive induction chemotherapy.
* Participants starting treatment with venetoclax in combination with azacytidine treated according to the Colombia label and who are not completed the first cycle (Cycle 28 days).

Exclusion Criteria:

- Participating in an interventional clinical trial within 30 days prior to Venetoclax treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed AML participants who are ineligible to intensive chemotherapy, that starting treatment with Venetoclax in combination with azacytidine treated according to the Colombia label.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 18 months
  OS defined as the time from the date of start Venetoclax to the date of death from any cause.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Complete Remission (CR) | Up to 18 Months
  CR is defined according to the modified International Working Group (IWG) criteria for acute myeloid leukemia (AML) as no morphologic evidence of AML and absolute neutrophil count >=10^3 /μL (>=1.0 x 10^9 /L), platelets >=10^5 /μL (>=100 x 10^9 /L), red blood cell (RBC) transfusion independence, and bone marrow with <5% blasts. Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.
Percentage of Participants Achieving Complete Remission with Incomplete Marrow Recovery (Cri) | Up to 18 Months
  Cri is defined according to the modified IWG criteria for AML as all criteria as CR except for residual neutropenia <10^3 /μL (1,000/ μL), or thrombocytopenia <10^5 /μL (100,000/ μL). If all criteria for CR are meet except for RBC transfusion independence, this also fulfills Cri criteria.
Percentage of Participants Achieving Complete Remission with Incomplete Marrow Recovery (CRh) | Up to 18 Months
  CRh is defined according to the modified IWG criteria for AML as bone marrow with < 5% blasts and Peripheral blood neutrophil count of > 0.5 × 10^3 /μL and Peripheral blood platelet count of > 0.5 × 10^5 /μL and 1-week (>= 7 days) platelet transfusion-free period prior to the hematology lab collection.
Percentage of Participants Achieving Transfusion Independence | Up to 18 Months
  Transfusion ndependence is defined as a period of at least 56 days with no transfusion between the first dose of Venetoclax and the last dose of Venetoclax plus 30 days.
Event-Free Survival (EFS) | Up to 18 Months
  EFS defined as the time from the date of start Venetoclax to the date of morphologic relapse, progressive disease, resistant disease, treatment failure, or death from any cause.
Duration of Remission (DOR) | Up to 18 Months
  DOR defined as the time from the date of first CR, CRi or CRh to the earliest evidence of morphologic relapse, progressive disease, or death due to disease progression.
Duration of Treatment (DoT) | Up to 18 Months
  DoT defined as the time from the start of a therapy to the time of treatment discontinuation for any reason.
Percentage of participants with Adverse Events (AE) | Up to 18 Months
  AE, defined as any unfavorable medical event that is temporarily related to the use of the investigational product, which does not necessarily have a causal relationship with the investigational product.
Percentage of participants achieving Minimal Residual Disease (MRD) negativity | Up to 18 Months
  MRD negativity, defined as having less than 10^-3 residual blasts per leukocyte measured in the bone marrow.
Change in Health-Related Quality of Life (HRQOL) Score | Up to 18 Months
  HRQOL score, defined as a multidimensional construct defined as the subjective perception of the life as a whole, including physical, emotional, social, cognitive functions, disease symptoms and side effects of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- Colombia (7):
  - Hospital Pablo Tobón Uribe /ID# 248569, Medellín, Antioquia
  - Hospital Alma Mater de Antioquia /ID# 248562, Medellin, Bogota D.C.
  - Sociedad de Oncologia y Hematologia del Cesar /ID# 248615, Valledupar, Cesar Department
  - Coorp Hosp Juan Ciudad Sede Hospital Universitario Mayor Mederi /ID# 248570, Bogota DC, Cundinamarca
  - Clinica del Country /ID# 248430, Bogota, Cundinamarca
  - Fundación Santa Fé De Bogotá /ID# 248563, Bogotá, Cundinamarca
  - Fundación Valle Del Lili /ID# 248294, Cali, Valle del Cauca Department

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com